CLINICAL TRIAL: NCT01833039
Title: An Open-Label Treatment Use Protocol for Ibrutinib (PCI-32765) in Subjects With Relapsed or Refractory Mantle Cell Lymphoma
Brief Title: An Open Label Treatment Use Protocol for Ibrutinib in Subjects With Relapsed or Refractory Mantle Cell Lymphoma
Status: Approved for marketing | Type: Expanded Access
Sponsor: Janssen Biotech, Inc. (Industry)
Collaborators: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR101862; PCI-32765MCL4001 (Other: Janssen)
Record Dates: First submitted 2013-04-06; First posted 2013-04-16 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Relapsed or Refractory Mantle Cell Lymphoma
Keywords: Mantle Cell Lymphoma; Ibrutinib
MeSH Terms: conditions — Recurrence; Lymphoma, Mantle-Cell | interventions — ibrutinib

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Ibrutinib — Ibrutinib

SUMMARY:
The purpose of this study is to provide patients who have relapsed or refractory Mantle Cell Lymphoma (MCL) with early access to an investigational medication called ibrutinib (PCI-32765) and to collect safety information about the drug.

ELIGIBILITY:
Inclusion Criteria:

* Patients, 18 years of age and older, with Mantle Cell Lymphoma who have relapsed or refractory disease after prior therapy are eligible.

Exclusion Criteria:

* Patients eligible for enrollment in any other ongoing clinical study of ibrutinib are not eligible.
* Patients previously treated with ibrutinib are not eligible.
* Patients enrolled in another interventional clinical study with therapeutic intent are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (51):
- United States (44):
  - Phoenix, Arizona
  - Duarte, California
  - Los Angeles, California
  - Stanford, California
  - Denver, Colorado
  - Norwalk, Connecticut
  - Stamford, Connecticut
  - Washington D.C., District of Columbia
  - Miami Beach, Florida
  - Ocala, Florida
  - Orlando, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Springfield, Illinois
  - Goshen, Indiana
  - Sioux City, Iowa
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Metairie, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Worcester, Massachusetts
  - Detroit, Michigan
  - Rochester, Minnesota
  - Jefferson City, Missouri
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Omaha, Nebraska
  - Reno, Nevada
  - Hackensack, New Jersey
  - New Hyde Park, New York
  - New York, New York
  - Syracuse, New York
  - Cleveland, Ohio
  - Columbus, Ohio
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Watertown, South Dakota
  - Knoxville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - Burlington, Vermont
  - Morgantown, West Virginia
- Brazil (6):
  - Barretos
  - Florianópolis
  - Porto Alegre
  - Rio de Janeiro
  - Salvador
  - São Paulo
- San Juan, Puerto Rico

REFERENCES:
- See also: An Open-Label Treatment Use Protocol for Ibrutinib (PCI-32765) in Subjects With Relapsed or Refractory Mantle Cell Lymphoma — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=4530&filename=CR101862_CSR.pdf